CLINICAL TRIAL: NCT01378039
Title: Evaluation of Pathogenetic Mechanisms of Chronic Obstructive Pulmonary Diseases
Brief Title: Pathogenetic Mechanisms of Chronic Obstructive Pulmonary Diseases
Acronym: CAPTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Raimundas Sakalauskas, Professor, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 48/2004
Record Dates: First submitted 2011-05-31; First posted 2011-06-22 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: COPD; Asthma
Keywords: COPD; Asthma; Pathophysiology; Genetics; Phenotype; Treatment response
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Budesonide (Other): patients who gave their agreement were randomised to 3 months treatment with either inhaled budesonide (400 µg BD) or placebo
  Interventions: Drug: comparison of treatment effect on different markers

INTERVENTIONS:
Drug: comparison of treatment effect on different markers — inhaled budesonide (400 µg BD) or placebo BD
  Other Names: Budesonide

SUMMARY:
Asthma and chronic obstructive pulmonary disease(COPD) are common diseases, which tend to even increase in many countries. Both from a clinical and a pathophysiological point of view, this is an important issue. However, an understanding of the relationship between the complex array of cells and mediators involved in asthma and COPD is not yet fully dissected which makes difficult to find a specific and sensitive panel of biomarkers that can reflect intensity of these pathological processes and can help to predict the individual outcome.

DETAILED DESCRIPTION:
Objectives:

To evaluate the patterns of pathophysiology and genetic predisposition of COPD and asthma

Tasks:

To evaluate patients that respond to corticosteroids and those who do not

Compare the inflammatory markers:

* of COPD and asthma patients before and after treatment with inhaled glucocorticoids
* of COPD and asthma patients that respond to inhaled glucocorticoids and those who do not
* of nonsmokers and smokers asthma patients

To identify a small set of markers that can be used to predict corticosteroid-treatment response in patients with COPD.

To evaluate epigenetic factors

To compare gene mutation and polymorphism between study groups

To evaluate the relationship between genetic predisposition and pathophysiology, clinical symptoms

To evaluate the relationship between patterns of pathophysiology and clinical symptoms, lung function, quality of life in patients with chronic obstructive pulmonary diseases.

Visit 1 Written informed consent will be obtained

* A full medical, surgical, smoking, labour history. A physical examination will be performed
* Resting SaO2 will be measured, exhaled nitric oxide (FENO)
* Chest X-ray
* Patient will fulfil questionnaires
* Spirometry and bronchodilatation test
* Sputum induction and samples will be performed

Visit 2 • Blood samples for blood clotting test and immunological markers will be taken• Cough inhalation challenge

Visit 3

* Patient will be hospitalized to the Department of Pulmonology and Immunology
* Blood samples for genetic analysis will be taken
* Urinary samples will be taken• Methacholine challenge test Polysomnography
* Bronchoscopy (biopsy and BAL)
* Study drug administration

Visit 4 and 5

* Adverse events, COPD or asthma exacerbation, concomitant medications will be recorded, exhaled nitric oxide (FENO)
* Spirometry
* Patient will fulfil questionnaires
* Cough inhalation challenge

Visit 6

* Patient will fulfil questionnaires
* Spirometry and bronchodilatation test.
* Sputum induction and samples will be performed

Visit 7

• Blood samples for blood clotting test, immunological and genetic analysis will be taken• Cough inhalation challenge

Visit 8

* Patient will be hospitalized to the Department of Pulmonology and Immunology
* Urinary samples will be taken• Methacholine challenge test Polysomnography
* Bronchoscopy (biopsy and BAL)
* Further treatment administration

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 40-80 years inclusive.
* An established clinical history of COPD as defined by the GOLD guidelines.
* COPD patients with a baseline (pre-bronchodilator) FEV1 40-80% of predicted normal value; post-bronchodilator FEV1/FVC ratio ≤ 70% predicted.
* COPD patients with a smoking history (current or ex-smoker) of ≥10 pack years or those who have exposure to occupational dust and chemicals
* An established clinical history of asthma defined by the GINA recommendations.
* Subjects with out hypoxemia (all subjects must have an O2 saturation ≥88% on room air).

Control (healthy) subjects with baseline FEV1 >80% of predicted normal value

* A female is eligible to participate this study if she is of non-childbearing potential, or childbearing potential has a negative pregnancy test.
* Patients who did not use inhaled and oral corticosteroids 6 weeks and/or long acting bronchodilators 4 weeks before study.

Exclusion Criteria:

* There is a current respiratory disorder other than COPD and asthma (e.g. lung cancer, sarcoidosis, active tuberculosis etc.)
* Subjects who have had a COPD and asthma exacerbation or respiratory infection in the 4 weeks before Visit 1.
* Subjects with a chest X-ray indicating diagnosis other than COPD or asthma that might interfere with the study.
* Subjects who are unable to stop treatment with inhaled, and oral corticosteroids 6 weeks and/or long acting bronchodilators 4 weeks before study.
* Subjects receiving treatment with cromolyn sodium or nedocromil, oral beta2 - agonists, long acting anticholinergic, leucotriene modifiers
* Subjects who have had lung surgery.
* Subjects with bleeding diathesis.
* Subjects receiving treatment with long-term oxygen therapy.
* Subjects with serious, uncontrolled diseases those are uncontrolled on permitted therapy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in inflammatory cell numbers and inflammatory markers at 3 months | 3 months
  inflammatory cell numbers and inflammatory markers (cytokines, chemokines, etc.) in different tissue compartments (induced sputum, BAL, bronchial biopsies, blood) will be measured at baseline and 3 months after treatment with budesonide and compared with those from healthy subjects

SECONDARY OUTCOMES:
network analysis of quantitative proteomics of bronchial biopsies | 3 months
  pathways analysis will be performed on proteins obtained from bronchial biopsies from asthmatics and COPD patients at baseline and 3 months after treatment
change of lung function, exNO after 3 months of treatment | 3 months
  lung function measurements (spirometry, bronchial responsiveness measurement, capsaicin test) at baseline and 3 months after treatment with budesonide

CONTACTS AND LOCATIONS:
Overall Officials: Raimundas Sakalauskas, Prof., Principal Investigator — Kaunas University of Medicine

REFERENCES:
- [Derived] O'Neil SE, Sitkauskiene B, Babusyte A, Krisiukeniene A, Stravinskaite-Bieksiene K, Sakalauskas R, Sihlbom C, Ekerljung L, Carlsohn E, Lotvall J. Network analysis of quantitative proteomics on asthmatic bronchi: effects of inhaled glucocorticoid treatment. Respir Res. 2011 Sep 22;12(1):124. doi: 10.1186/1465-9921-12-124. PMID 21939520